CLINICAL TRIAL: NCT03815695
Title: A Randomized, Placebo-controlled, Double Blind, Single Ascending and Multiple Ascending Dose Study to Assess the Safety, Pharmacokinetics and Pharmacodynamics of FT-4202 in Healthy Volunteers and Sickle Cell Disease Patients
Brief Title: A SAD/MAD to Assess the Safety, PK/PD of FT-4202 in Healthy Volunteers and Sickle Cell Disease Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Forma Therapeutics, Inc. (Industry)
Collaborators: Medpace, Inc. (Industry)
Responsible Party: Sponsor
Organization: Novo Nordisk A/S (Industry)
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 4202-HVS-101
Record Dates: First submitted 2018-12-21; First posted 2019-01-24 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Healthy Volunteers; Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Intervention Model Description: Single ascending dose escalation and multiple ascending dose escalation study followed by an evaluation of food effects on absorption
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: randomized double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Single ascending dose cohorts in healthy subjects (Experimental): Healthy volunteer subject cohorts randomized 6:2 receiving a single dose of FT-4202 or placebo. The first cohort will receive 200 mg of FT-4202 or placebo. Dose escalation will occur if FT-4202 or placebo is tolerated. The maximum dose of FT-4202 or placebo will be 1500 mg.
  Interventions: Drug: FT-4202/Placebo
- Multiple ascending dose cohorts in healthy subjects (Experimental): Healthy volunteer subject cohorts randomized 9:3 to receive FT-4202 or placebo for 14 days continuous dosing. The first cohort will receive 100 mg of FT-4202 or placebo daily X 14 days. The maximum dose of FT-4202/placebo will be 600 mg FT-4202/placebo daily for 14 days.
  Interventions: Drug: FT-4202/Placebo
- Food Effect Cohort in healthy subjects (Experimental): Health Volunteer subject cohort of 10 subjects who will receive a single dose of FT-4202 with food and without food. Dose will be administered per the protocol defined dose.
  Interventions: Drug: FT-4202/Placebo
- Single ascending dose cohorts in SCD subjects (Experimental): Sickle cell disease subject cohort randomized 6:2 receiving a single dose of FT-4202 or placebo. The dose of FT-4202/placebo administered will be a dose that was found to be safe in healthy subjects.
  Interventions: Drug: FT-4202/Placebo
- Multiple ascending dose cohorts in SCD subjects (Experimental): Sickle cell disease subject cohorts randomized 9:3 to receive FT-4202 or placebo for 14 days continuous dosing. The dose of FT-4202/placebo administered will be a dose less than the maximum tolerable dose evaluated in MAD healthy volunteers.
  Interventions: Drug: FT-4202/Placebo
- 12-week dosing cohort in SCD subjects (Experimental): Sickle cell disease subjects cohort to receive up to 84 consecutive daily doses of open-label FT-4202. The dose of FT-4202 administered will not exceed the highest dose evaluated in the MAD SCD subject cohorts
  Interventions: Drug: FT-4202/Placebo

INTERVENTIONS:
Drug: FT-4202/Placebo — Participants will receive FT-4202/placebo and monitored for side effects while undergoing pharmacokinetics and pharmacodynamic studies
  Other Names: Etavopivat

SUMMARY:
FT-4202 is an oral small-molecule agonist of pyruvate kinase red blood cell isozyme (PKR) being developed for the treatment of hemolytic anemias. This initial study will characterize the safety, tolerability and the pharmacokinetics/pharmacodynamics (PK/PD) of a single ascending dose and multiple ascending doses of FT-4202 in the context of Phase 1 studies in healthy volunteers and sickle cell disease patients. The effects of food on the absorption of FT-4202 will also be evaluated in healthy volunteers.

DETAILED DESCRIPTION:
This is a first-in-human (FIH), Phase 1 study of FT-4202 that will characterize the safety, PK and PD of FT-4202 after a single dose and after repeated dosing first in healthy adult volunteers and then in adolescents or adults with sickle cell disease (SCD). Initially, a dose range of FT-4202 in single ascending dose (SAD) escalation cohorts will be explored in healthy subjects. Enrollment of healthy subjects into 2-week multiple ascending dose (MAD) escalation cohorts will be initiated once the safety and PK from at least two SAD cohorts is available to inform the doses for the 2-week MAD portion of the study. The MAD cohorts will then run in parallel to the single dose cohorts. A single dose cohort of healthy subjects is planned to understand food effects (FE) on the PK of FT-4202. After the SAD and FE studies in healthy subjects are completed, the safety, PK, and PD of a single dose of FT-4202 that was found to be safe in healthy subjects will then be evaluated in SCD subjects. Multiple dose studies in SCD subjects will then be initiated upon completion of MAD studies in healthy volunteers.

ELIGIBILITY:
SCD Key Inclusion Criteria:

* Must be between 12 and 65 years of age
* Previously diagnosed sickle cell disease (hemoglobin electrophoresis or genotype)
* Must have a minimum body weight of 40 kg (88 lbs) at the Screening Visit
* Must have the ability to understand and sign written informed consent (and assent where applicable), which must be obtained prior to any study-related procedures being completed
* All male and female patients of child bearing potential must agree to use medically accepted contraceptive regimen during study participation and for 90 days after last study drug administration
* Must be willing to abide by all study requirements and restrictions

SCD Key Exclusion Criteria:

* Had more than 6 episodes of vaso-occlusive crisis (VOC) within the past 12 months that required a hospital, emergency room, or clinic visit
* Had a least one episode of acute chest syndrome in the last 6 months
* Received any of the following approved therapies for use in SCD:

  * Hydroxurea (HU): excluded if started HU < 90 days prior to Day 1 of study treatment
  * Adakveo®: excluded if received an infusion within 14 days prior to Day 1 of study treatment
  * Oxbryta®: excluded if received a dose within 7 days prior to start of Day 1 of study treatment
* Received a red blood cell transfusion within 30 days of starting the study drug
* Hemoglobin < 7.0 g/dL or > 10.5 g/dL
* Unable to take and absorb oral medications

HEALTHY VOLUNTEER Inclusion Criteria: [Note: no longer recruiting subjects for this portion of the study]

* Subjects must be between 18 and 60 years of age
* Subjects must have the ability to understand and sign written informed consent, which must be obtained prior to any study-related procedures being completed
* Subjects must be in general good health, based upon the results of medical history, a physical examination, vital signs, laboratory profile, and a 12-lead ECG
* All males and females of child bearing potential must agree to use medically accepted contraceptive regimen during study participation and up to 90 days after
* Subjects must be willing to abide by all study requirements and restrictions

HEALTHY VOLUNTEER Exclusion Criteria: [Note: no longer recruiting subjects for this portion of the study]

* Evidence of clinically significant medical condition or other condition that might significantly interfere with the absorption, distribution, metabolism, or excretion of study drug, or place the subject at an unacceptable risk as a participant in this study
* History of clinically significant cardiac diseases including condition disturbances
* Abnormal hematologic, renal and liver function studies
* History of drug or alcohol abuse

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2018-12-11 (Actual); Primary Completion 2021-12-17 (Actual); Study Completion 2021-12-17 (Actual)

PRIMARY OUTCOMES:
Incidence, frequency, and severity of adverse events (AEs) per CTCAE v5.0 of a single ascending dose and multiple ascending doses of FT-4202 in adult healthy volunteers and SCD patients. | Up to 3 weeks of monitoring
Maximum observed plasma concentration (Cmax) | Up to 3 weeks of testing
Time to maximum observed plasma concentration (Tmax) | Up to 3 weeks of testing
Area under the plasma concentration-time curve from time zero until the 24-hour time point (AUC0-24) | Up to 3 weeks of testing
Area under the plasma concentration-time curve from time zero until the last quantifiable time point (AUC0-last) | Up to 3 weeks of testing
Area under the plasma concentration-time curve from time zero to infinity (AUC0-inf) | Up to 3 weeks of testing
Terminal elimination half-life (t1/2) | Up to 3 weeks of testing
Apparent clearance (CL/F) | Up to 3 weeks of testing
Apparent volume of distribution (Vd/F) | Up to 3 weeks of testing
Terminal disposition rate constant (Lz) | Up to 3 weeks of testing
Renal clearance (ClR) | Up to 3 weeks of testing

SECONDARY OUTCOMES:
Change from baseline in the levels of 2,3-diphosphoglycerate (DPG) and adenosine triphosphate (ATP) in the red blood cells (RBCs) of healthy volunteers and SCD patients after single and multiple doses of FT-4202. | Up to 3 weeks of testing
Model-based estimate of change from baseline QT interval corrected using Fridericia's correction formula (QTcF) and 90% confidence interval at the estimated Cmax after a single dose of FT-4202 in healthy volunteers | up to 7 days
Change from baseline heart rate after a single dose of FT-4202 in healthy volunteers | up to 7 days
Change from baseline PR after a single dose of FT-4202 in healthy volunteers | up to 7 days
Change from baseline QRS after a single dose of FT-4202 in healthy volunteers | up to 7 days
Change from baseline T-wave morphology after a single dose of FT-4202 in healthy volunteers | up to 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Cameron Trenor, MD, Study Director — Forma Therapeutics, Inc.
Locations (18):
- United States (18):
  - Woodland International Research Group (SCD subjects only), Little Rock, Arkansas
  - Collaborative Neuroscience Research, LLC (SCD subjects only), Long Beach, California
  - Pacific Research Partners (SCD subjects only), Oakland, California
  - UCSF Benioff Children's Hospital Oakland (SCD subjects only), Oakland, California
  - Advanced Pharma CR, LLC (SCD subjects only), Miami, Florida
  - Children's Healthcare of Atlanta (SCD subjects only), Atlanta, Georgia
  - Augusta University Medical Center (SCD subjects only), Augusta, Georgia
  - University of Illinois at Chicago (SCD subjects only), Chicago, Illinois
  - University of Maryland, Greenebaum Comprehensive Cancer Center (SCD subjects only), Baltimore, Maryland
  - Columbia University Medical Center (SCD subjects only), New York, New York
  - Levine Cancer Institute (SCD subjects only), Charlotte, North Carolina
  - Duke University Medical Center (SCD subjects only), Durham, North Carolina
  - University of Cincinnati Medical Center (SCD subjects only), Cincinnati, Ohio
  - Medpace Clinical Pharmacology Unit (Healthy Volunteers only), Cincinnati, Ohio
  - Cincinnati Children's Hospital Medical Center (SCD subjects only), Cincinnati, Ohio
  - Lynn Institute of Tulsa (SCD subjects only), Tulsa, Oklahoma
  - St. Jude Children's Research Hospital (SCD subjects only), Memphis, Tennessee
  - The University of Texas Health Science Center at Houston (SCD subjects only), Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Saraf SL, Hagar R, Idowu M, Osunkwo I, Cruz K, Kuypers FA, Brown RC, Geib J, Ribadeneira M, Schroeder P, Wu E, Forsyth S, Kelly PF, Kalfa TA, Telen MJ. Multicenter, phase 1 study of etavopivat (FT-4202) treatment for up to 12 weeks in patients with sickle cell disease. Blood Adv. 2024 Aug 27;8(16):4459-4475. doi: 10.1182/bloodadvances.2023012467. PMID 38640200
- [Derived] Forsyth S, Schroeder P, Geib J, Vrishabhendra L, Konstantinidis DG, LaSalvia K, Ribadeneira MD, Wu E, Kelly P, Kalfa TA. Safety, Pharmacokinetics, and Pharmacodynamics of Etavopivat (FT-4202), an Allosteric Activator of Pyruvate Kinase-R, in Healthy Adults: A Randomized, Placebo-Controlled, Double-Blind, First-in-Human Phase 1 Trial. Clin Pharmacol Drug Dev. 2022 May;11(5):654-665. doi: 10.1002/cpdd.1058. Epub 2022 Jan 12. PMID 35019238